CLINICAL TRIAL: NCT05885828
Title: The PRECISION-T2D Study: Precision Nutrition Study for Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Westlake University (Other)
Collaborators: The Third People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20230306ZJS002
Record Dates: First submitted 2023-03-23; First posted 2023-06-02 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
Keywords: N-of-1; plant-based diet; precision nutrition; continuous glucose monitoring; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Plant-Based

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plant-based diet (Experimental): Participants in this arm will be recommended to consume more fiber-rich foods, including whole grains, fruits, legumes and vegetables; to moderate their intake of fish, eggs and dairy products; and to avoid other animal products. All participants are instructed not to modify their exercise habits during the intervention period.
  Interventions: Other: White bread; Other: Whole wheat bread; Behavioral: Plant-based diet; Other: Follow-up visit every 1-2 years
- Conventional diabetic diet (Experimental): Participants in this arm will be recommended to have a diet following 2023 Chinese Diabetes Society guidelines. All participants are instructed not to modify their exercise habits during the intervention period.
  Interventions: Other: White bread; Other: Whole wheat bread; Other: Conventional diabetic diet; Other: Follow-up visit every 1-2 years

INTERVENTIONS:
Other: White bread — After wearing CGM on Day 1, participants will be provided with white bread (76-77g) and milk (250mL) for breakfast on Day 3, Day 4, Day 7, Day 8, Day 10, Day 12.
  Other Names: Breakfast A
Other: Whole wheat bread — After wearing CGM on Day 1, participants will be provided with wheat bread (85-86g) and milk (250mL) for breakfast on Day 2, Day 5, Day 6, Day 9, Day 11, Day 13.
  Other Names: Breakfast B
Behavioral: Plant-based diet — After wearing CGM on Day 1, participants will be asked to follow the plant-based diet in next 30 days.
  Arms: Plant-based diet
Other: Conventional diabetic diet — Volunteers will be asked to have a diet following 2023 Chinese Diabetes Society guidelines in next 30 days.
  Arms: Conventional diabetic diet
Other: Follow-up visit every 1-2 years — Participants will be visited every 1-2 years. At each visit, face-to-face interviews, specimen collection, anthropometric measurements, ultrasonography evaluation, laboratory tests, and multi-omics data will be conducted.

SUMMARY:
Food plays a crucial role in determining blood glucose levels, especially in people with type 2 diabetes. Precision nutrition, which involves individually tailored dietary interventions, can be a powerful tool in managing blood glucose levels in people with type 2 diabetes. Previous studies found that changes in gut microbiota resulted from the dietary intervention, such as plant-based diet, might subsequently lead to different glycemic responses, and then different health outcomes.

In this study, the investigators will characterize the blood glucose dynamics and gut microbiota of individuals with type 2 diabetes. They aim to assess the influence of plant-based diet on gut microbiota; they will also investigate the influence of gut microbiota on glycemic responses. Additionally, a series of individual N-of-1 trails will be integrated to compare the effects of a white bread breakfast and a whole wheat bread breakfast on glucose metabolism at the individual level.

DETAILED DESCRIPTION:
Choice of design: The study is a two-arm intervention study integrated with N-of-1 design.

Study population: Patients with type 2 diabetes.

Screening Assessment: Prospective participants will be selected based on the pre-defined inclusion and exclusion criteria. Recruitment will be done over the phone and via the social media.

Study duration: Each participant will take part in the study for a period of up to 1 month at baseline and have follow-up visits every 1-2 years.

Dietary intervention:

The PRECISION-T2D is a dietary intervention study. Upon admission, patients will be randomly assigned to two groups: plant-based diet and conventional diabetic diet. Throughout the hospitalization, all participants (n=200) will be given standardized meals. A dietitian will design the diet for both plant-based and conventional diabetic diet groups following 2023 Chinese Diabetes Society guidelines. Both diets comprised approximately 50-65% of energy from carbohydrates, 20-30% of energy from fat, 15-20% from protein. The plant-based diet had higher fiber content (25-30g) compared to the conventional diabetic diet (15-20g). Participants will be asked to consume the entire amount of food indicated for the standardized meals and to record any leftover food. All participants will be asked to track their meals, snacks and drinks with instructions on how to record their daily dietary information. Participants will also be advised not to modify their exercise habits during the course of the study. Upon discharge, Participants in the plant-based diet arm will be recommended to consume more fiber-rich foods, including whole grains, fruits, legumes and vegetables; to moderate their intake of fish, eggs and dairy products; and to avoid other animal products. Participants in the conventional diabetic diet arm will be recommended to have a diet following 2023 Chinese Diabetes Society guidelines. Individual N-of-1 trial design will be employed to all participants during day one to day twelve to compare the difference of postprandial glucose response to white bread or whole wheat bread. These two standard breakfasts will appear in pseudo-random order. During the participants' first baseline visit day, they will be asked to complete a baseline questionnaire to collect information on their lifestyle, dietary habits, history of medications, sleep quality and appetite. Anthropometric measurements, ultrasonography evaluation, and laboratory tests will be taken using standard protocols. Participants will then be asked to wear a continuous glucose monitor (CGM) for 14-day blood glucose monitoring, which will be done by a nurse. On day 14, participants will be asked to come in for a clinical visit where they will receive their CGM report and provide blood, saliva, urine and stool samples. On day 30, participants will be asked to come in for another clinical visit where they will provide blood, saliva, urine and stool samples.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes;
* Living in Hangzhou for at least five years;
* Have the willingness or ability to complete the intervention and sample collection

Exclusion Criteria:

* Mental and physical disability;
* Already is a vegetarian;
* Cancer and serious complications from type 2 diabetes, such as renal failure;
* Using insulin for more than 5 years;
* Unstable medical/medication status;
* Current alcohol or drug abuse;
* Taking antibiotics in the last three months

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2033-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiome profile | Day 1 and Day 31
  Shotgun metagenomic sequencing will be performed in stool samples.
Blood glucose profile | 2 weeks
  Real-time blood glucose fluctuations will be recorded using continuous glucose monitoring.

SECONDARY OUTCOMES:
Carotid plaque | At enrollment
  Grade carotid plaque using ultrasound.
Carotid intima-media thickness | At enrollment
  Measure of carotid intima-media thickness using ultrasound.
Number of participants with chronic kidney disease | Up to 10 years
  The serum creatine and urine creatine and protein will be measured and chronic kidney disease will be defined as an estimated glomerular filtration rate of <60 mL/min/1.73 m2 or and the presence of an elevated urine microalbumin/creatinine ratio. All cases will be verified by medical record review.
Cognitive function | Up to 10 years
  Cognitive function was measured by the Addenbrooke's Cognitive Examination-Revised (ACE-R). The original 26 components were combined to produce five subscores, 100 in total. The cutoff for dementia is 82-88/100.
Changes in fasting blood glucose | Day 1 and Day 31
  Fasting glucose will be examined in mmol/L.
Changes in fasting blood C-peptide | Day 1 and Day 31
  Fasting blood C-peptide will be examined in μg/L.
Changes in fasting blood HbA1c | Day 1 and Day 31
  Fasting blood HbA1c will be examined in %.
Changes in lipid metabolism | Day 1 and Day 31
  Triglyceride, cholesterol, high density lipoprotein cholesterol and low density lipoprotein cholesterol will be examined in mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Sheng Zheng, PhD, Principal Investigator — Westlake University
Locations (2):
- China (2):
  - Westlake University, Hangzhou, Zhejiang
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang